CLINICAL TRIAL: NCT05993676
Title: A Feasibility Trial of a Smartphone App to Support the Mental Health of UK Armed Forces Veterans (MeT4VeT)
Brief Title: MeT4VeT: Mental Health Toolkit for Military Veterans Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 583696; DPRF-19/20-11079 (Other: King's College London); 1074/MODREC/20 (Other: MODREC)
Record Dates: First submitted 2023-07-25; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-07

CONDITIONS: Mental Health Issue; Mental Health Wellness 1
Keywords: MeT4VeT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Sham Comparator): The control group received an app containing only signposting information about a range of statutory and third sector organisations that focused on veterans' mental health.
  Interventions: Behavioral: MeT4VeT mobile phone app: control
- Intervention (Active Comparator): The intervention group will receive a 'full' version of the app over the 1month trial period. The app consists of five core elements:
  1. Personas developed as an aide to the provision of psycho-education on how mental health difficulties might look in real life and to help participants identify symptoms of mental health difficulties in themselves.
  2. Daily life goals employing behavioural activation principles to encourage users to set a series of small tasks to help them achieve larger goals in different areas of their life e.g. work, family, physical health.
  3. Self-help tools to provide participants with a range of resources that they can use independently to help them manage symptoms of mental ill-health they may be experiencing.
  4. Tracking tools to allow users to monitor their own mental health and to see their progress across the elements of the app.
  5. A schedule of daily notifications to encourage participants to continue to engage with the app.
  Interventions: Behavioral: MeT4VeT mobile phone app: intervention

INTERVENTIONS:
Behavioral: MeT4VeT mobile phone app: control — The control/ sham comparator arm of the Mental Health Toolkit for Veterans (MeT4VeT) smart phone app contains only signposting information around support services available to military veterans
  Arms: Control
Behavioral: MeT4VeT mobile phone app: intervention — The Mental Health Toolkit for Veterans (MeT4VeT) smart phone app has been developed through careful and close collaboration with military veterans and key providers of veterans' mental healthcare services. The aim of this app is to provide both a degree of education to support military veterans' understanding of mental health and foster self-recognition and management of mental health symptoms whilst also encouraging those who need it to seek more formal support.
  The elements of the app have been chosen for inclusion as they represent the intersection between:
  1. Core components of cognitive behavioural therapy, the theoretical framework underwriting the app
  2. Behaviour change constructs
  Arms: Intervention

SUMMARY:
The proposed research involves the running of a feasibility trial to assess a smart phone app designed to support military veterans (as they transition out of the Armed Forces) experiencing mental health difficulties to monitor and manage their mental health, encouraging them to seek formal mental healthcare services if required. The trial will compare participants who are provided with the 'full' app (case group) with participants who receive a 'signposting only' feature free smartphone app, receiving the 'full' app 3months later once the research trial is over (control group).

The feasibility trial has two core aims:

1. To provide initial assessment of the practicality of testing the app Running of the feasibility trial will provide key information on the practical delivery of the app and measurement processes; enable an estimation of recruitment and retention of participants; as well as trialling a series of outcome measures. All participants taking part in the trial will be asked to complete a short (20minute) in app survey at three time points: baseline; baseline plus 1month; baseline plus 3months. This questionnaire will collect demographic information and employ a number of well-being and quality of life measures.
2. To provide initial feedback on the app The trial will qualitatively evaluate how those in the case group use the 'full' app (via collection of app usage data over a 1month trial period) and how easy to interact with, and potentially helpful, they consider the app might be (via a short 30minute telephone interview at the end of the 1month app trial period).

If the trial indicates that the app is acceptable and feasible then a full randomized control trial (subject to funding) will be run to assess the effectiveness of the app in supporting mental health. If proven acceptable then the app would be made freely available to all.

DETAILED DESCRIPTION:
In line with the Medical Research Council Complex Intervention Framework (Medical Research Council) the feasibility stage of developing an intervention is focused on three areas to assess the practical aspects of testing an intervention including:

* Testing procedures (technical app delivery; measurement processes)
* Estimating recruitment and retention (number of eligible/ interested participants; drop-out rates)
* Determining sample size (testing main outcome measures to determine appropriate sample size for a later randomised control trial)

In addition to this, the feasibility trial will provide feedback from participants on their reactions to the app including:

* Actual use of the app
* Satisfaction with the app
* How appropriate they believe the app to be
* Intent for continued use

This toolkit will provide those who participate in the research with an additional support tool which may help them to manage their own mental health during a potentially challenging period (as they transition out of the Armed Forces) and help them to identify a need for more formal support if required.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Own a smartphone
* Served at least 2 years in the UK Armed Forces
* Left the UK Armed Forces within the last 2 years
* Not currently undertaking formal mental health treatment (mental health therapy by a medical professional)
* Indicate a degree of mental health distress (assessed via a score of two or more on the GHQ-12

Exclusion Criteria:

* Those who display current suicidal ideation / self-harm

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 50 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Recruitment and retention: Number of interested participants | 5month recruitment period
  Calculate the total number of participants contacting the study team to express an interest in taking part in the study.
Recruitment and retention: Number of eligible participants | 5month recruitment period
  Calculate the total number of participants contacting the study team to express an interest in taking part in the study who are eligible to take part. Calculate this as a percentage of total number of interested participants.
Recruitment and retention: Response rate | 5month recruitment period
  Calculate the total number of eligible participants who went onto complete the consent form. Calculate this as a percentage of total number of eligible participants.
Recruitment and retention: One month follow up retention rates | Baseline plus 1 months (28 days), end of trial period
  Calculate the total number of participants enrolled onto the study who went onto complete the 1month follow up. Calculate this as a percentage of total number of enrolled participants.
Recruitment and retention 4: Three month follow up retention rates | Baseline plus 3 months (84 days)
  Calculate the total number of participants enrolled onto the study who went onto complete the 3month follow up. Calculate this as a percentage of total number of enrolled participants.
Recruitment and retention 5: Comparability of sample to MOD personnel | Baseline plus 3 months (84 days)
  Comparability of sample to Ministry of Defence statistics for major sub-groups of veterans (age, service branch, rank)
Trial procedures and outcome measures: Technical delivery | Baseline plus 1 months (28 days), end of trial period
  Evaluation of the technical delivery of the app was gained through gathering feedback from developers and participants, identifying any potential technical issues
Trial procedures and outcome measures: GHQ12 | Baseline plus 3 months (84 days)
  The General Health Questionnaire (GHQ-12) is a measure of common mental disorders such as anxiety and depression. It is a 12-item self-report questionnaire measured on a 4-point scale. Scores range from 0-12 with a score of 4 or more indicative of probable mental ill health.The difference between scores at baseline, day 28 (1month) and day 84 (3months) were calculated.
Trial procedures and outcome measures: PCL-C | Baseline plus 3 months (84 days)
  To evaluate symptoms of PTSD, the PTSD Checklist Civilian version (PCL-C) was used. It is a 17-item self-report questionnaire, measured on a 5-point scale from (1) not at all to (5) extremely. Scores range from 17 to 85, scores over 50 are indicative of possible PTSD. The difference between scores at baseline, day 28 (1month) and day 84 (3months) were calculated.
Trial procedures and outcome measures: Well-being | Baseline plus 3 months (84 days)
  Warwick Edinburgh Mental Well-being Scale (WEMWBS) measures mental well-being within the previous two weeks and is a 14-item self-report questionnaire measured on a 5-point scale from (1) none of the time to (5) all of the time. Scores range from 14 to 70 with higher scores indicative of greater mental well being. The difference between scores at baseline, day 28 (1month) and day 84 (3months) were calculated.
Trial procedures and outcome measures: WHO QOL-BREF | Baseline plus 3 months (84 days)
  Quality of life was assessed using the World Health Organization Quality of Life Assessment (WHOQOL-BREF), a 26-item self-report questionnaire divided into four domains: physical health; social relationships; psychological health; environmental health. It is measured on a 5-point scale, with a score of 0-100 calculated, where 100 equates to the best possible state of health. The difference between scores at baseline, day 28 (1month) and day 84 (3months) were calculated.
Trial procedures and outcome measures: Completion rates | Baseline plus 3 months (84 days)
  Examination of the feasibility of using the app to collection outcome measures was assessed via completion rates for each of the questionnaires (baseline; 1month follow up; 3month follow up)
Trial procedures and outcome measures: Sample size | Baseline plus 3 months (84 days)
  Sample size estimates for a future randomised control trial were assessed via changes in GHQ12 scores from baseline to 3month follow up.
Acceptability and usability: Usage | Baseline plus 1 month (28 days), end of initial trial period
  App usage data were collected from Google Analytics via Firebase (CA, USA) and included information such as the number of times the app was opened, the duration of each app use and the number of times specific sections of the app were used.
Acceptability and usability: MAUQ | Baseline plus 1 month (28 days), end of initial trial period
  The mHealth App Usability Questionnaire (MAUQ) was used to assess app usability at day 28. A 16 item version of the MAUQ of the self-report questionnaire was used, measured on a 7-point scale ranging from strongly disagree (1) to strongly agree (7). Participant responses were aggregated into overall usability and three other domains: ease of use and satisfaction, interface and functionality, and usefulness. The mean total score and the mean of each three domains were scored out of seven, with a score of four indicating a neutral response and higher scores indicating greater app usability.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Fear, Prof, Principal Investigator — King's College London; Sharon Stevelink, PhD, Principal Investigator — King's College London; Neil Greenberg, Prof, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parkes S, Croak B, Brooks SK, Stevelink SAM, Leightley D, Fear NT, Rafferty L, Greenberg N. Evaluating a Smartphone App (MeT4VeT) to Support the Mental Health of UK Armed Forces Veterans: Feasibility Randomized Controlled Trial. JMIR Ment Health. 2023 Aug 28;10:e46508. doi: 10.2196/46508. PMID 37639295